CLINICAL TRIAL: NCT05102253
Title: Transcutaneous Electrical Acupoint Stimulation (TEAS) and Dense Cranial Electroacupuncture Stimulation (DCEAS) for Psychiatric Sequelae and Related Biomarkers in Women Victims of Domestic Violence: a Randomized Controlled Trial
Brief Title: Acupuncture for Women Victims of Domestic Violence With Psychiatric Sequelae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 21-238
Record Dates: First submitted 2021-09-27; First posted 2021-11-01 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Depression; Domestic Violence; Psychiatric Disorder
Keywords: Depression; Domestic Violence; Psychiatric Sequelae; Acupuncture; Transcutaneous Electrical Acupoint Stimulation; TEAS; Dense Cranial Electroacupuncture Stimulation; DCEAS
MeSH Terms: conditions — Depression; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TEAS+DCEAS group (Experimental): Subjects assigned to TEAS+DCEAS group will receive TEAS+DCEAS in addition to routine care.
  Interventions: Procedure: Dense cranial electroacupuncture stimulation (DCEAS); Procedure: Transcutaneous electrical acupoint stimulation (TEAS)
- Wait-list control: Routine care group (Other): Subjects assigned to this group will continue their current routine care as usual.
  Interventions: Other: Wait-list control: Routine care

INTERVENTIONS:
Procedure: Dense cranial electroacupuncture stimulation (DCEAS) — DCEAS will be conducted for 2 sessions per week for 12 consecutive weeks. Electrical stimulation will be conducted on six pairs of forehead acupoints located on the frontal, parietal, and temporal scalp areas. The acupoints includes: Bai-Hui (GV20), Yin-Tang (EX-HN3), left and right Si-Shen-Cong (EX-HN1), Tou-Lin-Qi (GB15), Shuai-Gu (GB8), Tai-Yang (EX-HN5) and Tou-Wei (ST8).
  Disposable acupuncture needles will be inserted at a depth of 10-30 mm perpendicularly or obliquely into acupoints. Manual manipulation will be carried out for all acupoints to evoke needling sensation, followed by electrical stimulation. The stimulation intensity will be adjusted to a level at which patients felt most comfortable. Each session of treatment will last 30 min.
  Arms: TEAS+DCEAS group
Procedure: Transcutaneous electrical acupoint stimulation (TEAS) — TEAS will be done for 3 times per week for 12 consecutive weeks by participants at home. A training workshop will be conducted to instruct participants how to use TEAS stimulator. Briefly, TEAS will be delivered on the bilateral Nei-Guan (PC6), which is located on the anterior forearm, between the tendons of the palmaris longus and ﬂexor carpi radialis, at the junction of the distal sixth and proximal ﬁve sixths of the line connecting the middle points of the wrist and elbow crease.
  Constant current electrical impulses will be produced from a TEAS apparatus. Two electrode pads will be adhered onto the acupoint skin. The pulse amplitude will be adjusted to a level at which the perception of 'strong but comfortable' is achieved. Each session of treatment will last 30 min.
  Arms: TEAS+DCEAS group
Other: Wait-list control: Routine care — The routine care may include medications, advocacy intervention, and CBT. Post-trial treatment of TEAS+DCEAS will be offered to serve as a compensation for their participation.
  Arms: Wait-list control: Routine care group

SUMMARY:
This is an assessor-blinded, randomized controlled trial. A total of 110 women victims of domestic violence aged 18-65 years will be recruited from local community centers and domestic violence shelters (refugee centers). They will be randomly assigned to routine care combined with (n = 55) and without (n = 55) additional acupuncture (TEAS+DCEAS) for 12 weeks. Acupuncture therapy will be conducted with 2 DCEAS sessions at clinics and 3 TEAS sessions at home each week. The primary outcome is the Beck Depression Inventory II (BDI-II) for depression. Secondary outcomes include the 17-item Hamilton Depression Rating Scale (HAMD-17) for depression, Perceived Stress Scale (PSS) for stress, PTSD Check List-Civilian Version (PCL-C) for PTSD symptoms, Insomnia Severity Index (ISI) for sleep and 12-Item Short Form Survey (SF-12) for quality of life. Two 10-ml blood samples will be drawn respectively at baseline and at the end of 12-week study. A generalized linear mixed-effect model will be applied to compare treatment outcomes over time in the two groups and linear regression will be conducted to examine inter-correlations among clinical improvement and changes in biomarker levels.

DETAILED DESCRIPTION:
Domestic violence, also referred to as intimate partner violence which overwhelmingly targets women of marriage and cohabitation, is a serious global public health issue with nearly 30% of women who have experienced physical or sexual abuse by their intimate partners. In Hong Kong, there were 4.5%-10% of women who experienced a physical violence and approximately 14,000 domestic violence cases reported to police offices each year. Depression is the most common psychiatric sequela of domestic violence, with an average prevalence of 47.6% among women victims. Recent study has shown that 65.2% women survivors of intimate partner violence had mild to severe depression. Abused women also often experienced post-traumatic stress disorder (PTSD), anxiety, substance abuse, and even suicidal thoughts. Although multiple psychological therapies, such as advocacy, cognitive behavioral therapy (CBT), and empowerment are a mainstay of domestic violence victim interventions, a large portion of the victims could not achieve satisfactory response and have low acceptability for psychological interventions; this seems to be particularly apparent in Asian women. Psychological interventions may be limited to patients with mild symptoms with long-term engagement of professionals. The development of non-psychological therapies is therefore highly desired.

Acupuncture has been widely introduced into local clinics and hospitals of Hong Kong. Numerous studies have shown benefits and efficacy of acupuncture in the treatment of various psychiatric disorders, including depression and anxiety. In addition to traditional invasive acupuncture in which needles are inserted into acupoints on the body, a non-invasive acupuncture mode called transcutaneous electrical acupoint stimulation (TEAS) also has been used in the treatment of postoperative anxiety, depression, autism, smoking cessation, and drug dependence. Compared to invasive acupuncture, obviously, TEAS is more acceptable to patients and physicians as it is non-invasive, safer, and time-saving, without causing pain and needle phobia. Furthermore, TEAS can be performed by patients themselves at home. These suggest that a combination of invasive acupuncture and TEAS could serve as an effective and more acceptable intervention for the victims.

Over the past decade, the effectiveness of advocacy and Qigong interventions in domestic violence women victims has been evaluated. Also, investigators have completed a series of epidemiological and methodological studies on women victims of domestic violence in local and international communities, with over 30 related papers published. On the other hand, a novel acupuncture stimulation called dense cranial electroacupuncture stimulation (DCEAS) based on neuroanatomical rationales has been developed. In this mode, electrical stimulation is delivered on dense acupoints located on the forehead innervated by the trigeminal nerve. Several clinical trials have confirmed the benefits and efficacy of DCEAS in patients with depression, obsessive-compulsive disorder (OCD), and neuropsychiatric sequelae of stroke. Moreover, two large-scale clinical trials have shown that patients with OCD and PTSD achieved an approximately 20% higher clinical remission rate on TEAS combined with CBT and/or antidepressants than those without TEAS. These results provide a solid foundation for further evaluation of the effectiveness of combining TEAS and DCEAS.

Besides, preliminary study has shown that several blood biomarkers were significantly correlated with the severity of depression and stress trauma. Determining relationships between potential biomarkers and the severity of psychiatric symptoms will lead people to better understand the pathogenesis of stress trauma and biochemical mechanisms of acupuncture effects.

These studies have led us to hypothesize that additional therapy with a combination of TEAS and DCEAS produces better outcomes than routine care alone in improving depression and other psychiatric sequelae of domestic violence; the therapeutic effects of acupuncture may be associated with the change of related biomarkers.

To test this hypothesis, an assessor-blinded, randomized controlled trial will be conducted to pursue the following two aims: (1) to compare the effectiveness of routine care with and without additional acupuncture in treating depression, stress, PTSD, insomnia symptoms, and quality of life of domestic violence women victims; and (2) to determine baseline-to-endpoint changes in levels of different blood biomarkers and their correlations with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Chinese women aged 18-65 years;
* have experienced domestic violence in the previous two years, confirmed with the Abuse Assessment Screen (AAS) Screen Questionnaire; and
* are currently experiencing a major depressive episode according to the criteria defined in the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5), with a BDI-II score of at least 14.

Exclusion Criteria:

* have serious medical conditions that may limit their participation in TEAS or DCEAS;
* have a history of brain injury or surgery;
* pregnancy or lactation;
* have investigational drug treatment in the previous 6 months;
* have heart pacemaker or other metal/electrical devices implanted in the body; or
* have severe needle phobia.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Beck Depression Inventory-II (BDI-II) | Baseline, Week 3, Week 6 and Week 12
  BDI-II is used to measure the severity of depression. Higher scores indicate greater severity. Assessments will be conducted at baseline, week 3, week 6 and week 12.

SECONDARY OUTCOMES:
Changes in 17-item Hamilton Depression Rating Scale (HAMD-17) | Baseline, Week 3, Week 6 and Week 12
  HAMD-17 is used to measure the severity of depression. Higher scores indicate greater severity. Assessments will be conducted at baseline, week 3, week 6 and week 12.
Changes in Perceived Stress Scale (PSS) | Baseline, Week 3, Week 6 and Week 12
  Stress is measured using PSS. Assessments will be conducted at baseline, week 3, week 6 and week 12.
Changes in PTSD Check List-Civilian Version (PCL-C) | Baseline, Week 3, Week 6 and Week 12
  PTSD symptoms are measured using PCL-C. Assessments will be conducted at baseline, week 3, week 6 and week 12.
Changes in Insomnia Severity Index (ISI) | Baseline, Week 3, Week 6 and Week 12
  Severity of insomnia are measured using ISI. Assessments will be conducted at baseline, week 3, week 6 and week 12.
Changes in Pittsburgh Sleep Quality Index (PSQI) | Baseline, Week 3, Week 6 and Week 12
  Sleep quality is assessed using PSQI. Assessments will be conducted at baseline, week 3, week 6 and week 12.
Changes in 12-Item Short Form Survey (SF-12) | Baseline, Week 3, Week 6 and Week 12
  Quality of life is measured using SF-12. Assessments will be conducted at baseline, week 3, week 6 and week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin Zhang, MMed, PhD, Principal Investigator — School of Chinese Medicine, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tiwari A, Fong DY, Yuen KH, Yuk H, Pang P, Humphreys J, Bullock L. Effect of an advocacy intervention on mental health in Chinese women survivors of intimate partner violence: a randomized controlled trial. JAMA. 2010 Aug 4;304(5):536-43. doi: 10.1001/jama.2010.1052. PMID 20682933
- [Background] Cheung DST, Deng W, Tsao SW, Ho RTH, Chan CLW, Fong DYT, Chau PH, Hong AWL, Fung HYKY, Ma JLC, Tiwari AFY. Effect of a Qigong Intervention on Telomerase Activity and Mental Health in Chinese Women Survivors of Intimate Partner Violence: A Randomized Clinical Trial. JAMA Netw Open. 2019 Jan 4;2(1):e186967. doi: 10.1001/jamanetworkopen.2018.6967. PMID 30646209
- [Background] Hackett S, McWhirter PT, Lesher S. The Therapeutic Efficacy of Domestic Violence Victim Interventions. Trauma Violence Abuse. 2016 Apr;17(2):123-32. doi: 10.1177/1524838014566720. Epub 2015 Jan 22. PMID 25612799
- [Background] Sun KS, Lam TP, Piterman L, Lam KF, Tang WS, Kwok KW, Chan HY, Wu D, Tiwari A. Management of Domestic Violence by Primary Care Physicians in Hong Kong: Association With Barriers, Attitudes, Training, and Practice Background. J Interpers Violence. 2021 Oct;36(19-20):9623-9647. doi: 10.1177/0886260519869067. Epub 2019 Aug 17. PMID 31423927
- [Background] Amorim D, Amado J, Brito I, Fiuza SM, Amorim N, Costeira C, Machado J. Acupuncture and electroacupuncture for anxiety disorders: A systematic review of the clinical research. Complement Ther Clin Pract. 2018 May;31:31-37. doi: 10.1016/j.ctcp.2018.01.008. Epub 2018 Jan 31. PMID 29705474
- [Background] World Health Organization. Global and regional estimates of violence against women: prevalence and health effects of intimate partner violence and non-partner sexual violence. Geneva: World Health Organization, 2013.
- [Background] Smith CA, Armour M, Lee MS, Wang LQ, Hay PJ. Acupuncture for depression. Cochrane Database Syst Rev. 2018 Mar 4;3(3):CD004046. doi: 10.1002/14651858.CD004046.pub4. PMID 29502347
- [Background] Feng B, Zhang Y, Luo LY, Wu JY, Yang SJ, Zhang N, Tan QR, Wang HN, Ge N, Ning F, Zheng ZL, Zhu RM, Qian MC, Chen ZY, Zhang ZJ. Transcutaneous electrical acupoint stimulation for post-traumatic stress disorder: Assessor-blinded, randomized controlled study. Psychiatry Clin Neurosci. 2019 Apr;73(4):179-186. doi: 10.1111/pcn.12810. Epub 2019 Jan 22. PMID 30565342
- [Background] Feng B, Zhang ZJ, Zhu RM, Yuan GZ, Luo LY, McAlonan GM, Xu FZ, Chen J, Liu LY, Lv YY, Wong HK, Zhang Y, Zhu LX. Transcutaneous electrical acupoint stimulation as an adjunct therapy for obsessive-compulsive disorder: A randomized controlled study. J Psychiatr Res. 2016 Sep;80:30-37. doi: 10.1016/j.jpsychires.2016.05.015. Epub 2016 May 28. PMID 27281260
- [Background] Greene MC, Rees S, Likindikoki S, Bonz AG, Joscelyne A, Kaysen D, Nixon RDV, Njau T, Tankink MTA, Tiwari A, Ventevogel P, Mbwambo JKK, Tol WA. Developing an integrated intervention to address intimate partner violence and psychological distress in Congolese refugee women in Tanzania. Confl Health. 2019 Aug 17;13:38. doi: 10.1186/s13031-019-0222-0. eCollection 2019. PMID 31428190
- [Background] Wong JY, Tiwari A, Fong DY, Bullock L. A Cross-Cultural Understanding of Depression Among Abused Women. Violence Against Women. 2016 Oct;22(11):1371-96. doi: 10.1177/1077801215624791. Epub 2016 Jan 21. PMID 26796779
- [Background] Zhang ZJ, Wang XM, McAlonan GM. Neural acupuncture unit: a new concept for interpreting effects and mechanisms of acupuncture. Evid Based Complement Alternat Med. 2012;2012:429412. doi: 10.1155/2012/429412. Epub 2012 Mar 8. PMID 22474503
- [Background] Zhang ZJ, Ng R, Man SC, Li TY, Wong W, Tan QR, Wong HK, Chung KF, Wong MT, Tsang WK, Yip KC, Ziea E, Wong VT. Dense cranial electroacupuncture stimulation for major depressive disorder--a single-blind, randomized, controlled study. PLoS One. 2012;7(1):e29651. doi: 10.1371/journal.pone.0029651. Epub 2012 Jan 6. PMID 22238631
- [Background] Zhang ZJ, Zhao H, Jin GX, Man SC, Wang YS, Wang Y, Wang HR, Li MH, Yam LL, Qin ZS, Yu KT, Wu J, Ng FB, Ziea TE, Rong PJ. Assessor- and participant-blinded, randomized controlled trial of dense cranial electroacupuncture stimulation plus body acupuncture for neuropsychiatric sequelae of stroke. Psychiatry Clin Neurosci. 2020 Mar;74(3):183-190. doi: 10.1111/pcn.12959. Epub 2019 Dec 20. PMID 31747095
- [Background] Zhang ZJ, Wang XY, Tan QR, Jin GX, Yao SM. Electroacupuncture for refractory obsessive-compulsive disorder: a pilot waitlist-controlled trial. J Nerv Ment Dis. 2009 Aug;197(8):619-22. doi: 10.1097/NMD.0b013e3181b05fd1. PMID 19684500
- [Background] Man SC, Hung BH, Ng RM, Yu XC, Cheung H, Fung MP, Li LS, Leung KP, Leung KP, Tsang KW, Ziea E, Wong VT, Zhang ZJ. A pilot controlled trial of a combination of dense cranial electroacupuncture stimulation and body acupuncture for post-stroke depression. BMC Complement Altern Med. 2014 Jul 19;14:255. doi: 10.1186/1472-6882-14-255. PMID 25038733
- [Background] Zhang ZJ, Wang D, Man SC, Ng R, McAlonan GM, Wong HK, Wong W, Lee J, Tan QR. Platelet 5-HT(1A) receptor correlates with major depressive disorder in drug-free patients. Prog Neuropsychopharmacol Biol Psychiatry. 2014 Aug 4;53:74-9. doi: 10.1016/j.pnpbp.2014.03.004. Epub 2014 Mar 20. PMID 24657886
- [Background] Malki K, Keers R, Tosto MG, Lourdusamy A, Carboni L, Domenici E, Uher R, McGuffin P, Schalkwyk LC. The endogenous and reactive depression subtypes revisited: integrative animal and human studies implicate multiple distinct molecular mechanisms underlying major depressive disorder. BMC Med. 2014 May 7;12:73. doi: 10.1186/1741-7015-12-73. PMID 24886127
- [Background] https://www.edb.gov.hk/attachment/tc/teacher/student-guidance-discipline-services/lecture-notes/lecture-notes-201718/20180103_Identification_and_ intervention.pdf
- [Derived] Yang S, Tiwari A, Cheung DST, Cheng CPW, Chan MY, Chen H, Zhang ZJ. Electrical acupoint stimulation for psychiatric sequelae in women victims of domestic violence: study protocol for an assessor-blind randomized controlled trial. BMC Complement Med Ther. 2025 Sep 1;25(1):316. doi: 10.1186/s12906-025-05033-3. PMID 40890795